CLINICAL TRIAL: NCT06011369
Title: A Prospective , Controlled, Randomized Multi-center Study on the Usefulness of Fluorescence in Thyroid Surgery
Brief Title: Study of Usefulness of Fluorescence in Thiroid Surgery
Acronym: ECA_SPAFLUO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMIB-SPAFLUO
Record Dates: First submitted 2023-08-01; First posted 2023-08-25 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Thyroid Surgery
MeSH Terms: interventions — Fluorescence

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE, CONTROLLED, RANDOMIZED
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluorescence in thyroid surgery (Experimental): Patients undergoing thyroid surgery with cervical fluorescence.
  Interventions: Procedure: Fluorescence in thyroid surgery
- No Fluorescence in thyroid surgery (No Intervention): patients undergoing thyroid surgery without cervical fluorescence.

INTERVENTIONS:
Procedure: Fluorescence in thyroid surgery — Fluorescence in thyroid surgery
  Arms: Fluorescence in thyroid surgery

SUMMARY:
In thyroid surgery, the identification and preservation of the parathyroid glands and their vascularization is essential to avoid postoperative hypoparathyroidism. In this sense, fluorescence technology with autofluorescence (AF) can help us avoid this post-surgical complication. This study aims to determine the advantages offered by fluorescence in thyroid surgery, taking into account various clinical variables.

For this, a randomized study is proposed in patients undergoing thyroid surgery with and without cervical fluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Total thyroidectomy with/without lymph node dissection
* Signature of informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Hemithyroidectomy
* Reintervention of thyroid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Type of surgery performed | Up to 12 months.
  total thyroidectomy/hemithyroidectomy; lymphadenectomy
Number of parathyroid glands identified before the use of AF (Autofluorescence) | Up to 12 months.
  Gland count
Number and location of parathyroid glands identified with the use of FA (Autofluorescence) | Up to 12 months.
  Gland count
Quantification of each parathyroid gland with AF(Autofluorescence) | Up to 12 months.
  (two determinations in the same parathyroid gland, in total, eight determinations of the parathyroid glands parathyroid, and three determinations in the thyroid gland, the last being in a nodule if it'd exist
Number of glands accidentally removed. | Up to 12 months.
  Gland count
Number of autotransplanted glands. | Up to 12 months.
  Gland count
Surgical time. | Up to 12 months.
  Hours of surgery
Number of previous thyroidectomies performed with FA (Autofluorescence)(learning curve) | Up to 12 months.
  Number of surgeries using autofluorescence
Concentration of PTH and calcium corrected by albumin and/or ionic | 4, 24 Hours
  Value in analytics
Concentration of PTH and calcium corrected by albumin and/or ionic | 6,12 Months
  Value in analytics

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Febrero, MD, Principal Investigator — HCUVA
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No